CLINICAL TRIAL: NCT01393574
Title: Comparing Treatment With Melatonin to Treatment With Stimulants (Methylphenidate) in Children With Attention Deficit Hyperactivity Disorder and Sleep Difficulties
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: principal investigator: Dr. Amir Ytzhak, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 83/11
Record Dates: First submitted 2011-07-12; First posted 2011-07-13 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Attention Deficit Hyperactivity Disorder; Sleep Onset Insomnia
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Melatonin; Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melatonin treatment (Experimental): Treatment with Melatonin before sleep for 1 month - 3 mg for body weight <40kg, 6mg for body weight >40kg
  Interventions: Drug: Melatonin
- Stimulants treatment (Active Comparator): Treatment with Methylphenidate with a formulary and dose as decided by the treating neurologist, for 1 month.
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Melatonin — 3 mg for body weight <40kg, 6 mg for body weight >40kg, once a day 30-60 minutes before sleep
  Arms: Melatonin treatment
Drug: Methylphenidate — Drug formulary and dose will be decided by the treating neurologist from the available options in Israel (as would be given if not participating in the trial)
  Other Names: Ritalin; Ritalin SR; Ritalin LA; Concerta
  Arms: Stimulants treatment

SUMMARY:
The study hypothesis is that some children with Attention-Deficit-Hyperactivity-Disorder (ADHD) who also have sleep onset difficulties will improve with Melatonin treatment to an extent similar to that of stimulants treatment.

In order to check this hypothesis children with a new ADHD diagnosis who also have sleep difficulties will be treated with either Melatonin or with stimulants (Methylphenidate) for one month. The main outcome will be improvement of the ADHD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* children 6-18 years old with a new ADHD diagnosis who are candidates for treatment with stimulants
* Also they suffer from sleep onset insomnia or difficult awakening

Exclusion Criteria:

* Drug treatment for ADHD or for sleep problems in the last 6 months
* Any other chronic medical treatment
* Sleep disorder requiring a different treatment
* Asthma in the last 2 years

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
ADHD symptoms improvement | a month
  ADHD symptoms improvement - a clinical judgement based on history from the patient and parents, and from the teacher report

SECONDARY OUTCOMES:
Sleep difficulties improvement | 1 month
  Sleep difficulties improvement - clinical judgement based on history from the patient and parents and from a sleep diary.

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Haroffeh Medical Center, Zeriffin, Israel